CLINICAL TRIAL: NCT01660737
Title: Observational Study With PASCALLERG ® in Patients With Hay Fever
Status: Completed | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 180A12PALL
Record Dates: First submitted 2012-08-01; First posted 2012-08-09 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Hay Fever
Keywords: Hay fever; Pascallerg
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PASCALLERG® tablets in patients with hay fever: Patients with lactose intolerance and / or chromium hypersensitivity are excluded from the observational study.

SUMMARY:
The aim of this observational study is to document the therapeutic use of PASCALLERG ® for hay fever. Based on the survey is a decrease in disease-specific symptoms when taking PASCALLERG ® over a period of 4 weeks will be documented. In addition to the compatibility can be assessed.

DETAILED DESCRIPTION:
There are documented male and female patients over the age of one year who suffer from hay fever. The traetment time is about a period of 4 weeks with PASCALLERG® tablets.

ELIGIBILITY:
Inclusion Criteria:

* hay fever

Exclusion Criteria:

* Lactose intolerance and / or
* Chromium hypersensitivity

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients from natural practioners and doctors from Germany
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jennifer Lebert, Giessen, Germany

REFERENCES:
- [Derived] Trompetter I, Lebert J, Weiss G. Homeopathic complex remedy in the treatment of allergic rhinitis: results of a prospective, multicenter observational study. Forsch Komplementmed. 2015;22(1):18-23. doi: 10.1159/000375244. Epub 2015 Feb 9. PMID 25824400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Started | 123
Completed | 123
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 84
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.00 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 58
Region of Enrollment [Number; unit: participants]
  Germany | 123

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pascallerg
Description: Request of Efficacy using a 4-stage scale (very good efficacy, good efficacy, moderate efficacy, no efficacy)
Time Frame: appr. 4 weeks after baseline (after appr. 4 weeks of treatment)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 123
participants
  Very good efficacy (symptoms complete decline) | 60
  Good efficacy (symptoms clearly improved) | 44
  Moderate efficacy (smptoms slightly improved) | 15
  No efficacy (symptoms unchanged o worsend) | 2
  No data available | 2

2. Primary Outcome: Tolerability of Pascallerg
Description: Request of Tolerability using a 2-stage scale (very good tolerability, bad tolerability)
Time Frame: app. 4 weeks after baseline (treatment app. for 4 weeks)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 123
participants
  Very good | 122
  Bad tolerability | 1

3. Secondary Outcome: Numerical Rating Scale Well Beeing (Pre- Post)
Description: Influence of allergy on the general well-being (scale from 0-no influence to 10 strong influence)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 115
participants
  improved | 109
  unchanged | 4
  detoriorated | 2

4. Secondary Outcome: Change of Symptom Dry Eyes (Pre- Post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 45
participants
  improved | 36
  unchanged | 9
  deteriorated | 0

5. Secondary Outcome: Change of Symptom Itching Eyes (Pre- Post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 101
participants
  improved | 87
  unchanged | 10
  deteriorated | 4

6. Secondary Outcome: Change of Symptom Burning Eyes (Pre-post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 76
participants
  improved | 68
  unchanged | 6
  deteriorated | 2

7. Secondary Outcome: Change of Symptom Bronchial Complaints (Pre-post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 54
participants
  improved | 44
  unchanged | 7
  deterioreated | 3

8. Secondary Outcome: Change of Symptom Sneezing (Pre-post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 107
participants
  improved | 87
  unchanged | 13
  deteriorated | 7

9. Secondary Outcome: Change of Symptom Rhinitis (Pre-post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 102
participants
  improved | 89
  unchanged | 8
  deteriorated | 5

10. Secondary Outcome: Change of Symtom Fatigue / Tiredness
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 93
participants
  improved | 77
  unchanged | 11
  deteriorated | 5

11. Secondary Outcome: Change of Symptom Headache (Pre-post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 53
participants
  improved | 38
  unchanged | 15
  deteriorated | 0

12. Secondary Outcome: Change of Symptom Tearing Eyes (Pre-post)
Description: Request Scale (0=not present, 1=mild, 2=moderate, 3=strong)
Time Frame: Change from Baseline (before treatment; week 0) to last visit (end of observation- approx. 4 weeks after baseline)
Measure: Number; unit: participants
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Number analyzed (Participants) | 82
participants
  improved | 70
  unchanged | 7
  deteriorated | 5

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | PASCALLERG® Tablets in Patients With Hay Fever
Serious Adverse Events (participants affected / at risk) | 0/123
Other Adverse Events (participants affected / at risk) | 1/123
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PASCALLERG® Tablets in Patients With Hay Fever (N=123)
rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No